CLINICAL TRIAL: NCT04282408
Title: Experimental Evaluation of Back Braces for the Treatment of Spinal Deformity Produced With 3D Printing Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: National Research Council of Italy - IPCB (Unknown); Orthopedic Center "Biomedica Su Misura" (Brescia, Italy) (Unknown); Orthopedic Center "Labsan" (Lecco, Italy) (Unknown); Politecnico di Milano - DIG Department (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GIP673
Record Dates: First submitted 2020-02-11; First posted 2020-02-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Adolescent Idiopathic Scoliosis; Osteogenesis Imperfecta
Keywords: scoliosis; spinal deformity
MeSH Terms: conditions — Osteogenesis Imperfecta; Scoliosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Group treated with 3D printed brace
  Interventions: Device: Scoliosis back brace

INTERVENTIONS:
Device: Scoliosis back brace — The patients will use the traditional brace, if not already in use, for 2 weeks and then they will wear a 3D printed back brace for the following 2 weeks. Both the braces will be worn for the amount of hours per day prescribed by the physician.

SUMMARY:
The proposed investigation is a pilot study that involves pediatric patients affected by spinal deformity (Adolescent Idiopathic Scoliosis and Osteogenesis Imperfecta).

The main goal is to evaluate the acceptability, the safety and the overall satisfaction of the patients wearing the back braces produced with an innovative methodology using 3D printers, compared to the current braces manufactured with a production model based on thermoforming, that has well-established clinical efficacy.

ELIGIBILITY:
Inclusion Criteria for Adolescent Idiopathic Scoliosis:

* ages 6 to 17 years;
* lumbar or thoracolumbar scoliosis;
* measured rib hump greater than 5 degrees with scoliometer;
* Cobb angle, measured on frontal X-ray images, within 15 and 30 degrees.

Inclusion Criteria for Osteogenesis Imperfecta:

* ages 3 to 17 years;
* vertebral pain and/or vertebral deformity with typical double-concave lenses shape and/or deformity in frontal or sagittal planes assessed with clinical traction, deflection or derotational tests.

Exclusion Criteria:

* skin allergies;
* behavioural and psychiatric problems (e.g., emotional problems, anxiety, panic);
* chest dimensions beyond printing limits (i.e., maximum diameter 35 cm and maximum height 60 cm).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Comfort and safety evaluation by using surveys | Comparison between traditional and 3D printed brace after 2 weeks of usage of each.
  The patients have to fill in ad hoc surveys with open and closed questions about their personal experience with the traditional brace only and after the use of the 3D printed brace. In the closed questions they will have to mark a score from 1 to 7, where higher values correspond to better outcome.

SECONDARY OUTCOMES:
Production process time evaluation | The design and manufacturing will take place in the first 2 weeks between the first and the second visit.
  The innovative process will be analysed by recording the time for each phase, from the geometry acquisition with 3D scanning to the delivery of the final 3D printed brace.
Material amount evaluation | The meaasurements will take place immediately after the brace is removed from the printer and right before delivering the brace to the patient in its final layout.
  The production process will be also analyzed in term of amount of material used: both for the final product and for the part wasted in building supports.
Stability assessment with and without braces measured by sway area | After 2 weeks of treatment with the 3D printed brace.
  Data are collected with an inertial sensor while performing the following task: maintaining a static standing position for 1 minute (3 repetitions), both with and without the braces.
Gait symmetry metric with and without braces | After 2 weeks of treatment with the 3D printed brace.
  Data are collected with an inertial sensor while performing the following task: Timed Up and Go (TUG) test (3 repetitions).

OTHER OUTCOMES:
Thermal distribution on the braces | After 2 weeks of treatment with the thermoformed and the 3D printed brace.
  The subjects will be acquired with both the braces (thermoformed and 3D printed) and without using a thermal camera in order to evaluate the temperature distribution and analyse the differences among the different conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy

REFERENCES:
- [Derived] Costantini S, Redaelli DF, Fraschini P, Biffi E, Storm FA. On mobility and gait in scoliosis patients: a comparison of conventional and 3D-printed braces during an instrumented timed-up and go test. BMC Musculoskelet Disord. 2025 Jan 27;26(1):86. doi: 10.1186/s12891-025-08311-w. PMID 39871223